CLINICAL TRIAL: NCT00045006
Title: Phase I Clinical Trial of Oral Suberoylanilide Hydroxamic Acid - SAHA (MSK390) in Patients With Advanced Solid Tumors and Hematologic Malignancies
Brief Title: Suberoylanilide Hydroxamic Acid in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: MSKCC-01021; CDR0000256306 (Registry Identifier: PDQ (Physician Data Query)); ATON-0101; NCI-G02-2099
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2003-10

CONDITIONS: Cancer
Keywords: acute undifferentiated leukemia; de novo myelodysplastic syndromes; borderline ovarian surface epithelial-stromal tumor; ovarian sarcoma; ovarian stromal cancer; previously treated myelodysplastic syndromes; prolymphocytic leukemia; recurrent adult Hodgkin lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent bladder cancer; recurrent breast cancer; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent metastatic squamous neck cancer with occult primary; recurrent mycosis fungoides/Sezary syndrome; recurrent non-small cell lung cancer; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; recurrent prostate cancer; recurrent renal cell cancer; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; stage III multiple myeloma; stage III mycosis fungoides/Sezary syndrome; stage III ovarian germ cell tumor; stage IV mycosis fungoides/Sezary syndrome; stage IV ovarian germ cell tumor; unspecified adult solid tumor, protocol specific; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage III bladder cancer; stage IV bladder cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; stage III oropharyngeal cancer; stage IV oropharyngeal cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; stage III prostate cancer; stage IV prostate cancer; stage III renal cell cancer; stage IV renal cell cancer; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent salivary gland cancer; stage IV salivary gland cancer; stage III salivary gland cancer; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent basal cell carcinoma of the lip; stage III basal cell carcinoma of the lip; stage IV basal cell carcinoma of the lip; recurrent mucoepidermoid carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; recurrent verrucous carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; male breast cancer
MeSH Terms: conditions — Neoplasms; Leukemia, Biphenotypic, Acute; Leukemia, Prolymphocytic; Hodgkin Disease; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Urinary Bladder Neoplasms; Breast Neoplasms; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Mycosis Fungoides; Sezary Syndrome; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial; Prostatic Neoplasms; Carcinoma, Renal Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Multiple Myeloma; Oropharyngeal Neoplasms; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Breast Neoplasms, Male | interventions — Vorinostat

INTERVENTIONS:
Drug: vorinostat

SUMMARY:
RATIONALE: Suberoylanilide hydroxamic acid may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth.

PURPOSE: Phase I trial to study the effectiveness of suberoylanilide hydroxamic acid in treating patients who have advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of suberoylanilide hydroxamic acid in patients with advanced solid tumors or hematologic malignancies.
* Evaluate the pharmacokinetic profile of this drug in these patients.
* Determine the effects of this drug on absorption in the fasting and non-fasting states in these patients.
* Determine any anti-tumor effects of this drug in these patients.
* Correlate clinical outcomes with histone acetylation in circulating mononuclear cells and tumor biopsy samples in patients treated with this drug.

OUTLINE: This is a dose-escalation study. Patients are stratified according to disease (solid tumor vs multiple myeloma or lymphoma vs leukemia or myelodysplastic syndromes).

The initial 15-20 patients (in the solid tumor or multiple myeloma or lymphoma stratum) receive suberoylanilide hydroxamic acid (SAHA) IV over 2 hours on day 1 of week 0 and then orally once or twice daily beginning on day 1 of week 1. All remaining patients receive oral SAHA once or twice daily beginning on day 1 of week 1. Courses repeat every 4 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.

In each stratum, cohorts of 3-6 patients receive escalating doses of SAHA until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed monthly for resolution of adverse events.

PROJECTED ACCRUAL: A maximum of 114 patients (42 with solid tumors, 36 with lymphoma or multiple myeloma, and 36 with leukemia or myelodysplastic syndromes) will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following diagnoses:

  * Histologically confirmed advanced primary or metastatic solid tumor, including, but not limited to, the following:

    * Androgen-independent prostate cancer
    * Breast cancer
    * Ovarian cancer
    * Head and neck cancer
    * Non-small cell lung cancer
    * Bladder cancer
    * Kidney cancer
  * Diagnosis of lymphoma, multiple myeloma, leukemia, or myelodysplastic syndromes (MDS), including, but not limited to, the following:

    * Intermediate-grade or follicular non-Hodgkin's lymphoma
    * Hodgkin's lymphoma
* Patients with lymphoma or multiple myeloma must be ineligible for peripheral blood stem cell transplantation
* For patients with solid tumors (except prostate cancer):

  * Disease progression based on development of new lesions or an increase in pre-existing lesions
  * Biochemical marker increase must not be sole criterion for disease progression
* For prostate cancer patients only:

  * Disease progression based on rising prostate-specific antigen (PSA) values, transaxial imaging, or radionuclide scans
  * Increase in disease-related symptoms must not be sole manifestation of progression
  * Patients receiving an antiandrogen as part of first-line hormonal therapy must show disease progression off of the antiandrogen prior to study
  * Biochemical progression (at least 25% increase over range of values) defined as 1 of the following:

    * Rising PSA documented by at least 3 consecutive measurements obtained at least 1 week apart
    * Rising PSA documented by at least 2 consecutive measurements obtained more than 1 month apart
  * PSA at least 4 ng/mL

    * Testosterone no greater than 50 ng/mL
    * If no prior orchiectomy, must maintain castrate levels of testosterone
* Disease must be refractory to standard therapy or for which no curative therapy exists
* No active CNS or epidural tumors
* Hormone receptor status:

  * Not specified NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,500/mm^3
* Platelet count at least 100,000/mm^3 (patients with solid tumors)
* Platelet count greater than 25,000/mm^3 (patients with hematologic malignancy)
* Absolute neutrophil count at least 500/mm^3 (patients with hematologic malignancy)

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 3 times ULN
* PT no greater than 15 seconds

Renal

* Creatinine no greater than 2.0 mg/dL

Cardiovascular

* No New York Heart Association class III or IV heart disease

Pulmonary

* No severe debilitating pulmonary disease

Other

* No infection requiring IV antibiotics
* No other severe medical problems that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* At least 4 weeks since prior chemotherapy

Endocrine therapy

* See Disease Characteristics
* At least 4 weeks since prior ketoconazole
* At least 2 weeks since prior steroids for patients with lymphoma
* Concurrent gonadotropin-releasing hormone analogs or diethylstilbestrol to maintain castrate levels of testosterone allowed for prostate cancer patients
* No concurrent ketoconazole

Radiotherapy

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy to sole measurable lesion

Surgery

* See Disease Characteristics
* No concurrent surgery

Other

* Recovered from all prior therapy
* At least 4 weeks since prior palliative therapy for solid tumor patients with progressive metastatic disease (if present)
* At least 4 weeks since prior investigational anticancer therapeutic drugs
* At least 2 weeks since prior conventional cytotoxic therapy for patients with leukemia or MDS
* At least 4 weeks since prior investigational therapy for patients with leukemia or MDS
* No other concurrent investigational drugs
* No other concurrent anticancer agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-07; Primary Completion 2005-12 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William K. Kelly, DO, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States